CLINICAL TRIAL: NCT06327542
Title: Group-based Integrative Pain Management: A Multi-level Approach to Address Intersectional Stigma and Social Isolation in Diverse Primary Care Safety Net Patients With Chronic Pain
Brief Title: Group-based Integrative Pain Management in Primary Care Safety Net Clinics
Acronym: IPMP+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 22-37078B; 4R33MD018333 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: health equity; integrative health; nonpharmacologic pain management; stigma; social isolation; primary care; group medical visits
MeSH Terms: conditions — Chronic Pain; Social Stigma; Social Isolation

STUDY DESIGN:
Intervention Model Description: 2x2 factorial trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): Participants will receive care as usual provided through their primary care providers. Usual care includes medical diagnostic evaluation, analgesic drug therapies, recommendations for physical activity, and sometimes referral to specialist physicians or physical therapy. Usual care was chosen as a comparison arm for this study because it is practical and clinically relevant. Participants randomized to usual care will be put on a waitlist and can access group acupuncture or IGMV after their final study visit.
- Group Acupuncture (Experimental): Participants randomized to acupuncture will receive 12 weeks of acupuncture treatments delivered in a group setting, dosing similar to prior research. Acupuncture point selection and other treatment details will follow responsive manualization, a protocol developed for the largest clinical trial of group acupuncture to date. A licensed acupuncturist experienced with administering group acupuncture treatments will determine each participant's traditional Chinese medicine diagnosis and administer 8-10 acupuncture needles on distal points of participant's body (below the knees, from the elbows to the hands, and on the head). Duration of assessment, needle placement and retention will be 30-45 minutes. Details of acupuncture treatments (e.g., frequency and duration, traditional Chinese medicine diagnosis, number of needles and points used) will be documented in electronic health records.
  Interventions: Other: Group Acupuncture
- Integrative Group Medical Visits (IGMV) (Experimental): IGMV will consist of a 12-week program that provides education on the biopsychosocial model of pain and multimodal treatments; physical movement; mindfulness training; and peer support. Non-pharmacologic approaches are based on guidelines on chronic pain management; feedback of experts, staff, and patients; and feasibility with the greatest potential to benefit participants. Participants will receive a binder with educational materials.
  Interventions: Other: Integrative Group Medical Visits
- Group Acupuncture and IGMV (Experimental): Both group acupuncture and IGMV. Along with usual care, participants will be offered weekly group acupuncture treatments and integrative group medical visits as described above.
  Interventions: Other: Group Acupuncture; Other: Integrative Group Medical Visits

INTERVENTIONS:
Other: Group Acupuncture — Acupuncture will be delivered in a group setting, in a common space with multiple reclining chairs. Acupuncture treatments will include a 10-15 minute diagnostic intake with the acupuncturist, followed by administration of acupuncture needles retained for 20-40 minutes. Acupuncture points will be selected based on a treatment manual developed for the study. All treatments will be administered using sterile, disposable, surgical stainless steel acupuncture needles.
  Arms: Group Acupuncture; Group Acupuncture and IGMV
Other: Integrative Group Medical Visits — IGMV sessions will be weekly for 90-120 minutes in a group meeting space. Sessions will start with a "check-in" where participants can share their emotions, thoughts, hopes, and fears related to their health and pain and provide updates since the last session. Group sessions will be led by a primary care provider and a health educator and will include psychosocial support, tools for pain self-management, and psychoeducation for pain management. Invited experts will provide information on educational topics, including neurobiology of pain, medication safety, and connections between mood and pain, as well as participatory activities such as therapeutic movement or mindfulness practice.
  Arms: Group Acupuncture and IGMV; Integrative Group Medical Visits (IGMV)

SUMMARY:
Socioeconomically disadvantaged populations have a high prevalence of chronic pain, exacerbated by social isolation, intersectional stigma, and disparities in pain assessment and treatment options. Effective interventions using a multilevel, biopsychosocial approach are needed to decrease the unequal burden of pain. The proposed study will test group-based integrative models of pain management in primary care safety net clinics to improve pain care for racially and ethnically diverse low-income patients.

DETAILED DESCRIPTION:
Background: The proposed study seeks to address chronic pain disparities in racially diverse, socioeconomically disadvantaged individuals by optimizing multimodal pain management provided in primary care safety net clinics. Multilevel barriers exist in primary care settings where socioeconomically disadvantaged patients are most often treated. Lack of access to multimodal and nonpharmacologic care at the organizational level alongside provider bias and other forms of discrimination at the interpersonal level contribute to unequal assessment, treatment, and quality of pain care. Stigmatization cross-cuts all levels and is closely linked with social isolation common among individuals with chronic pain. Group-based models are a promising multilevel approach to increase access to non-pharmacologic therapies, address time constraints that contribute to disparities in pain care, improve patient-clinician communication, and provide social support among safety net patients with chronic pain.

Methods: This study uses mixed methods and a pragmatic 2x2 randomized factorial trial to test two group-based models: integrative group medical visits (IGMV) and group acupuncture. In collaboration with primary care safety net clinics, the investigators will recruit and randomize 360 participants to (1) IGMV, (2) group acupuncture, (3) both, or (4) neither (usual care, waitlist control). IGMV includes pain education, social and behavioral support, and mind-body approaches (meditation, yoga). Participants randomized to IGMV will initiate groups once enough participants for a cohort have enrolled (8-12 patients). Group acupuncture uses responsive manualization, allowing for a standardized yet individualized treatment. Participants randomized to group acupuncture will initiate 12 weeks of treatment once baseline is completed. Study participants will be asked to complete a total of 3 assessments: a pre-test (baseline), post-test at 3-months, and final follow-up 6 months after baseline.

The investigators will test the hypotheses that compared with usual care, group acupuncture and IGMV improve pain outcomes among racially and ethnically diverse, low-income patients with chronic pain. Our co-primary outcomes of interest are changes in pain impact from baseline to three months (a composite score of pain intensity, pain interference, and physical function) and social support in chronic pain.

Secondary outcomes include: pain interference, pain intensity, physical function, depression, anxiety, sleep, social functioning, global physical, mental, and social well-being using National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS®) measures. The investigators will also examine intervention effects on social isolation, internalized stigma of chronic pain, and experiences of discrimination. The investigators will also conduct focus groups and semi-structured interviews to further understand patient experiences with pain management, patient-clinician relationships, and clinical care in primary care safety net settings.

Significance: Multilevel approaches are needed to advance health equity in pain management. The proposed study will contribute to knowledge of group-based integrative pain management co-located in primary care to address disparities in pain care for socioeconomically vulnerable populations. The study receives support from the Helping to End Addiction Long-term® (HEAL) Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18
* Fluency in English or Spanish
* Panelled to a primary care provider at one of the study clinics
* Diagnosis of chronic pain (> 3 months)
* Had a primary care visit for chronic pain within the past six months
* Ability to provide a phone number
* Able to participate in groups
* Intent to be available for up to 24 weeks

Exclusion Criteria:

* Received group-based pain management in the past 3 months
* Received acupuncture treatment for pain in the past 3 months
* Active cancer treatment
* Inability to provide informed consent due to mental illness or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain impact measured as a composite score of pain intensity, pain interference, and physical function. | Baseline, 12 weeks, and 24 weeks
  Self-reported pain impact will be measured as a composite score of pain intensity, pain interference and physical function. These scores are summed to create Pain Impact, which ranges from 3-50, with higher scores indicating greater impact of pain on one's life, capturing overall day-to-day physical function, the impact of pain on ability to do regular life tasks, and the intensity of pain experienced.
Change in Social support and Pain Questionnaire (SPQ) | Baseline, 12 weeks, and 24 weeks
  Social Support in Chronic Pain will be measured using Van Der Lugts' 6-item Social support and Pain Questionnaire (SPQ). Total scores range from 0 to 24, with higher scores indicating greater levels of social support.

SECONDARY OUTCOMES:
Change in average pain intensity on the 0-10 numeric rating scale | Baseline, 12 weeks, and 24 weeks
  Pain intensity in the past 7 days will be measured on the numeric rating scale (NRS), the score ranges from 0-10, with zero indicating no pain and 10 indicating the worst pain imaginable.
Self-reported pain interference will be measured using the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) scale. Total t-scores range from 0 to 100, with higher scores indicating greater levels of pain interference. | Baseline, 12 weeks, and 24 weeks
  Change in pain interference on the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 8a survey
Change in physical function on the 6-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 6b | Baseline, 12 weeks, and 24 weeks
  Self-reported physical function will be measured using the 6-item NIH PROMIS Physical Function Short Form 6b. Total t-scores range from 0 to 100, with higher scores indicating more optimal levels of physical function.
Change in Internalized Stigma of Chronic Pain (ISCP) survey | Baseline, 12 weeks, and 24 weeks
  Internalized Stigma of Chronic pain will be measured using the 21-item ISCP, with subscales for enacted and internalized chronic pain stigma. Total scores range from 1 to 4, with high scores indicating greater levels of internalized stigma.
Change in social isolation on the 8-item NIH Patient Reported Outcomes Measurement Information System (PROMIS) Social Isolation Short Form 8a | Baseline, 12 weeks, and 24 weeks
  Self-reported social isolation will be measured using the 8-item PROMIS Social Isolation Short Form 8a scale. Total t-scores range from 0 to 100, with higher scores indicating greater levels of social isolation.
Change in pain self efficacy on the Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 12 weeks, and 24 weeks
  Pain self efficacy will be measured on a 10 item measure Pain Self-Efficacy Questionnaire (PSEQ) developed by Nicholas. Total scores range from 0 to 60 with higher scores indicating stronger self-efficacy beliefs.
Change in pain catastrophizing on the Pain Catastrophizing Scale (PCS) 6-item short form | Baseline, 12 weeks, and 24 weeks
  Pain catastrophizing will be measured using the Pain Catastrophizing Scale 6-item short form. Total scores range from 0 to 24, with higher scores indicating greater levels of pain catastrophizing.
Change in depressive symptoms on the Patient Health Questionnaire (PHQ-9) | Baseline, 12 weeks, and 24 weeks
  Self-reported depressive symptoms will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Total scores range from 0 to 27, with higher scores indicating greater levels of depressive symptoms.
Change in anxiety on the Generalized Anxiety Disorder survey (GAD-2) | Baseline, 12 weeks, and 24 weeks
  Self-reported anxiety will be measured using the 2-item Generalized Anxiety (GAD-2). Total scores range from 0 to 6, with higher scores indicating greater levels of anxiety.
Patient belief about treatment efficacy on the Patient Global Impression of Change (PGIC) | 12 weeks and 24 weeks
  Patient belief about treatment efficacy will be measured using a single item patient global impression of change (PGIC). Total score rates from 0 (very much improved) to 6 (very much worse).
Change in health-related quality of life on NIH Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale | Baseline, 12 weeks, and 24 weeks
  Health-related quality of life will be measured using the 4-item NIH PROMIS Global Health Scale which measures sleep disturbance, social functioning, global physical, mental, and social well-being. Total t-scores range from 0 to 100, with higher scores indicating greater well-being.
Change in experiences of discrimination in healthcare | Baseline, 12 weeks, and 24 weeks
  Experiences of discrimination in healthcare will be measured using the 7-item Perceived Discrimination in Healthcare Scale. Total scores range from 0 to 28, with high scores indicating greater levels of perceived discrimination in healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chao, DrPH, MPA, Principal Investigator — University of California, San Francisco
Locations (1):
- Tom Waddell Urban Health Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will comply with NIH Helping to End Addiction Long term (HEAL) policies on data sharing, which will include depositing deidentified data in a data repository.
Supporting Information: Study Protocol, ICF
Time Frame: To be determined based on NIH HEAL policies
Access Criteria: Access to trial IPD can be requested by qualified researchers, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.